CLINICAL TRIAL: NCT05000242
Title: West Hertfordshire Inflammatory Bowel Disease Technology Study
Acronym: WHITS
Status: Active, not recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: West Hertfordshire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20/LO/0349
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Disease; Ulcerative Colitis; Crohns Disease; Artificial Intelligence; Endoscopy; Pathology; Radiology
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective and prospective, observational, non-interventional, cohort study to develop quantitative metrics from tools used as standard of care when diagnosing, assessing and monitoring patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
Inflammatory bowel disease is a chronic inflammatory disease of the gastrointestinal tract that is without cure. It comprises two main disorders: Crohn's disease and ulcerative colitis. These conditions can lead to debilitating symptoms of abdominal pain, weight loss, diarrhoea and rectal bleeding.

The incidence of inflammatory bowel disease is increasing worldwide and is increasingly considered an emerging global disease. The prevalence of inflammatory bowel disease is currently the highest in North America and Western Europe and up to 600,000 people in the United Kingdom are thought to be affected.

The diagnosis and monitoring of inflammatory bowel disease is based on clinical, endoscopic, radiological and histological features. Endoscopy, is considered the current gold standard in inflammatory bowel disease with newer techniques being developed. There are however limitations to these methods, especially regarding the inter and intra observer variability in assessing the validated scoring systems used from the gold standard modalities.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 16 or over
* Patients with known or suspected Inflammatory Bowel Disease scheduled to undergo clinical, endoscopic or radiological assessment
* Patients with known Inflammatory Bowel Disease under ongoing clinical monitoring, who have previously undergone clinical, endoscopic or radiological assessments.
* Participant willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Participant who is, or suspects that they are, pregnant at the time of assessment
* Any other cause, including significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This research aims to develop digital tools specifically to aid patients with:
  1. Left sided, extensive or Pan-colonic Ulcerative colitis, undergoing flexible sigmoidoscopy or colonoscopy
  2. PaIleocolonic or colonic Crohn's disease undergoing flexible sigmoidoscopy or colonoscopy
  3. Post-operative Crohn's disease undergoing colonoscopic assessment of surgical anastomosis
  4. Ileal Crohn's disease undertaking or having previously undertaken small bowel CT or MRI
  5. Crohn's disease with perianal disease undergoing or having previously undertaking pelvic MRI
  6. A previous admission for acute severe ulcerative colitis
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Development and presentation of computer generated metrics derived from endoscopic videos. | 24 months
  To develop quantitative metrics from computational modelling of endoscopic, histological and radiological data by comparing clinical scores for inflammatory bowel disease between computer and human generated metrics to aid and improve assessment of inflammatory bowel disease.
Development and presentation of computer - generated metrics derived from histology slides. | 24 months
  To develop quantitative metrics from computational modelling of endoscopic, histological and radiological data by comparing clinical scores for inflammatory bowel disease between computer and human generated metrics to aid and improve assessment of inflammatory bowel disease.
Development and presentation of computer generated metrics derived from Magnetic Resonance Elastography/ Computerised Tomography Enterography / Magnetic Resonance Imaging Pelvis scans. | 24 months
  To develop quantitative metrics from computational modelling of endoscopic, histological and radiological data by comparing clinical scores for inflammatory bowel disease between computer and human generated metrics to aid and improve assessment of inflammatory bowel disease.

SECONDARY OUTCOMES:
The relation between human and computer generated metrics will be assessed using Cohen's Kappa (k) and correlation coefficients (Pearson's/Spearman's). | 24 months
  To determine whether quantitative metrics produced from digitised versions of inflammatory bowel disease investigatory tools accurately correspond to current standard care endoscopic, radiological and histological assessment in inflammatory bowel disease.
Bland Altman analysis (bias, slope of bias, Limits of Agreement, the corresponding 95% Confidence Interval) and Inter-Class Correlation coefficients will be reported to estimate agreement between variables as endpoints for repeatability/reproducibility. | 24 months
  To compare repeatability and reproducibility of humangenerated and computer-generated metrics
Statistical performance of computer diagnostic tools compared to clinical diagnoses: sensitivity, specificity, Area Under Receiver Operating Curve, predictive positive/negative value, survival curves with respect to clinical diagnosis/disease severity. | 24 months
  To determine the diagnostic and prognostic ability of the novel quantitative metrics to predict/diagnose clinical outcome data in addition to patient response to therapies and surgeries. This will be derived from historical and prospective endoscopic, imaging, clinical and histopathological data.
Performance of metrics will be assessed using Cohen's Kappa (k) and Inter-Class Correlation coefficient. | 24 months
  To determine inter-observer and intra-observer variability in human-generated and computer generated metrics

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Landy, Study Chair — West Hertfordshire Trust
Locations (1):
- West Hertfordhsire Teaching Hospitals NHS Trust, Watford, Hertfordshire, United Kingdom